CLINICAL TRIAL: NCT03933839
Title: Internet-Based Pain Coping Skills Training (PainCOACH) for Patients With Lupus
Brief Title: Internet-Based Pain Coping Skills Training for Patients With Lupus
Acronym: PainCOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0600
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PainCOACH (Experimental): This group will take part in an 8-week pain coping skills training (PCST) intervention.
  Interventions: Behavioral: PainCOACH
- Wait List Control (No Intervention): The other group will be the wait list group and will receive the pain CST program after completing all study measures.

INTERVENTIONS:
Behavioral: PainCOACH — PainCOACH is an eight-week, automated, internet-based training in specific pain coping skills (such as progressive muscle relaxation, pleasant imagery and activity pacing), and guided practice with each skill.
  Arms: PainCOACH

SUMMARY:
This is a pilot study of an automated, internet-based pain coping skills training (PCST) program, PainCOACH.

DETAILED DESCRIPTION:
Background and Significance: Systemic lupus erythematosus (SLE) is a chronic autoimmune disease that impacts multiple organ systems. SLE results in a variety of challenging symptoms, including flare-ups and periods of remission that are unpredictable, and it is a complex disease to manage clinically. Because of these factors, SLE often has a major impact on patients' quality of life. Notably, SLE is often associated with pain, fatigue, emotional symptoms like anxiety and depression, and disability. Because of the relatively young average age of SLE onset, many patients must navigate these challenges while maintaining work and / or caring for young children.

Prior studies show that greater use of adaptive coping strategies and greater self-efficacy for coping with SLE-related symptoms are associated with better physical and psychological outcomes. Conversely, maladaptive coping behaviors, particularly pain catastrophizing (e.g., focusing on and exaggerating the threat of pain and negatively evaluating one's ability to deal with pain), are associated with poorer SLE outcomes. Importantly, many studies in other rheumatic conditions have shown that pain coping skills training (PCST) programs can improve coping patterns, as well as physical and psychological health outcomes. However, there have been no trials of PCST among individuals with SLE, who face a unique set of disease-related challenges and are overall younger than patients with many other rheumatic conditions. Delivery of PCST programs to patients with SLE could have a tremendous impact on outcomes and quality of life, but this evidence base needs to be established, including adaptations of current PCST programs that may be important specifically for patients with SLE. Therefore, the objective of this project is to conduct a pilot study of an automated, internet-based PCST program, PainCOACH, that has been shown to improve multiple key outcomes among patients with osteoarthritis

Study Aims: This project has three specific aims: 1) Evaluate the feasibility and acceptability of PainCOACH among patients with SLE. 2) Obtain a preliminary assessment of the efficacy of PainCOACH (relative to a wait list control group) for improving pain interference and other key outcomes among patients with SLE 3) Determine appropriate adaptations to PainCOACH for patients with SLE.

Study Description: Investigators will conduct a randomized pilot study, with N=60 patients age >= 18 years with physician diagnosis of systemic lupus erythematosus (SLE), equally allocated to PainCOACH and a wait list control group that will be offered PainCOACH after completion of the 9 week follow-up assessment. This design will allow a between-group comparison as well as collection of acceptability data from the control group following their completion of PainCOACH. Outcomes will be assessed at baseline and at about 9 week follow-up as PainCOACH is designed for delivery over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosis of Systemic lupus erythematosus (SLE)

Exclusion Criteria:

* significant memory loss
* active psychosis or substance abuse
* neuropsychiatric SLE
* severe hearing impairment
* inability to speak English
* pregnant or planning to become pregnant in the next 3 months
* current participation in another SLE-related trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 9 weeks in PROMIS Pain Interference Score | Baseline and 9 weeks
  PROMIS Pain Interference (Short Form 6a) includes 6 items assessing self-reported consequences of pain across aspects of life including social, cognitive, emotional, physical and recreational activities rated on a Likert scale of 1 (not at all) to 5 (very much). Scores are converted to t-scores and higher scores indicate greater pain interference. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like pain interference, a T-score of 60 is one SD worse than average. By comparison, a pain interference T-score of 40 is one SD better than average.

SECONDARY OUTCOMES:
Change from Baseline to 9 weeks in PROMIS-29 Score | Baseline and 9 weeks
  PROMIS-29 includes 29 items covering 7 domains of self-reported health rated on a 5 point Likert scale. There is also one 11-point rating scale for pain intensity. Norm-based scores have been calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population (standard deviation = 10).High scores represent more of the domain being measured. Thus, on symptom oriented domains of PROMIS-29 (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores represent worse symptomatology. On the function oriented domains (physical functioning and social role) higher scores represent better functioning.
Change from Baseline to 9 weeks in Coping Strategies Questionnaire (CSQ) Score | Baseline and 9 weeks
  CSQ includes 48 items that assess 6 cognitive domains (Catastrophizing, Diverting Attention, Ignoring Sensations, Coping Self-Statements, Reinterpreting Pain Sensations, Praying-Hoping) and 1 behavioral domain (Increasing Behavioral Activities). Each domain includes 6 items, and participants rate the frequency of their use of specific coping strategies on a 7-point Likert scale from 0 ("Never do that") to 6 ("Always do that"). A Total Coping Attempts score was created, which includes 5 cognitive domains and 1 behavioral domain but excludes the Catastrophizing domain, similar to prior studies. Total range is 252, with higher scores indicating more coping attempts.
Change from Baseline to 9 weeks in LupusPRO Score | Baseline and 9 weeks
  LupusPRO (v1.8) includes 43 items with domains of Lupus Symptoms, Lupus Medication, Physical Health, Emotional Health, Pain, Sleep, Procreation, Cognition, Body Image, Desires-Goals, Coping, Social Support and Satisfaction with Care rated on a 5 point Likert scale, where 0=None of the time/not applicable, 1= A little of the time, 2= Some of the time, 3=Most of the time, 4= All of the time, 5= Not applicable.
  Total scores measure health (HRQOL) and non-health related quality of life (Non HRQOL). Item scores are totaled for each domain item and the mean domain score is obtained by dividing the total score by the number of items in that domain. The mean raw domain score is transformed to scores ranging from 0 (worst QOL) to 100 (best QOL) by dividing by 4 (the number of Likert responses {5 responses} minus 1) and then multiplying by 100. Total HRQOL and N-HRQOL scores are obtained by averaging the transformed domain scores within each construct.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP
Time Frame: Data will become available following publication of primary and secondary outcomes, and data will be available until the study is closed with the local IRB.
Access Criteria: Data will be accessible following publication of study results and will be available until the study is closed with the local IRB.

REFERENCES:
- [Derived] Allen KD, Beauchamp T, Rini C, Keefe FJ, Bennell KL, Cleveland RJ, Grimm K, Huffman K, Hu DG, Santana A, Saxena Beem S, Walker J, Sheikh SZ. Pilot study of an internet-based pain coping skills training program for patients with systemic Lupus Erythematosus. BMC Rheumatol. 2021 Jun 17;5(1):20. doi: 10.1186/s41927-021-00191-6. PMID 34134788